CLINICAL TRIAL: NCT07192757
Title: Improving Speech in Noise Perception for Individuals With Age-related Hearing Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202500769
Record Dates: First submitted 2025-09-09; First posted 2025-09-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Presbycusis
Keywords: age-related hearing loss; taVNS; vagus nerve stimulation; presbycusis; hearing aids
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment A (Experimental): participants will receive low level electrical stimulation to the auricular branch of the vagus nerve during the sound in noise task
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- Treatment B (Active Comparator): Participants will receive stimulation to a control location
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — active electrical stimulation applied to the cymba conchae of the left ear
  Arms: Treatment A
Device: Sham Control — electrical stimulation applied to a location on the ear not innervated by the auricular vagus
  Arms: Treatment B

SUMMARY:
Hearing loss, especially for speech perception in the presence of noise, may lead older individuals to withdraw from social situations. While hearing aids help amplify sound and are useful in many situations, they can be ineffective in noisy contexts. The proposed pilot study will evaluate taVNS for improving speech in noise perception in adults with age-related hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Adults 55-80 years old
* Normal hearing or age-related hearing loss (with or without hearing aids)

Exclusion Criteria:

* History of traumatic brain injury or noise trauma
* Implanted medical devices (eg., pacemaker) or ferrous metal
* Known history of heart conditions
* Medications that impact neurotransmitters released by vagus nerve stimulation

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Speech in noise performance | 2 weeks
  Percent correct on a speech in noise perception task in participants receiving Treatment A compared to Treatment B

OTHER OUTCOMES:
Predictive value of audiometric testing | 2 weeks
  Scores on audiometric battery measures and how they differ in those receiving treatment A compared to those receiving treatment B
Predictive value of brain measures | 2 weeks
  Level of baseline GABA levels in primary auditory cortex prior to and following intervention in those receiving Treatment A compared to those receiving Treatment B

CONTACTS AND LOCATIONS:
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States